CLINICAL TRIAL: NCT05207397
Title: Lactate for Energy and Neurocognition
Acronym: LEAN
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: STUDY00144303; 1R01AG062548 (NIH)
Record Dates: First submitted 2021-08-09; First posted 2022-01-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Healthy Aging; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: Lactate clamp: After insertion of the catheters, and prior to isotope infusion, a background blood and breath sample (ParvoMedics TrueOne 2400) will be obtained. The investigator will then administer priming doses of 57.5 mg [13C3]lactate, 250 mg D2-glucose and 136 mg H13CO3- followed by continuous infusions of [13C3]lactate at 10 mg/min and D2-glucose at 2 mg/min. Along with the continuous isotope infusion the investigator will begin infusion of the Na-lactate at approximately 2.6mg/kg·min. Based upon readings from blood samples during the infusion, this rate will be adjusted as needed to maintain the target lactate concentration of approximately 4-5 mM. Blood samples will be drawn at 10, 20, 30, 45, 60, 75, 90 and 120 minutes, while breath samples will be collected at 60, 75, 90 and 120 minutes.
  Interventions: Other: Lactate infusion
- Mild Cognitive Impairment: Lactate clamp: After insertion of the catheters, and prior to isotope infusion, a background blood and breath sample (ParvoMedics TrueOne 2400) will be obtained. The investigator will then administer priming doses of 57.5 mg [13C3] lactate, 250 mg D2-glucose and 136 mg H13CO3- followed by continuous infusions of [13C3] lactate at 10 mg/min and D2-glucose at 2 mg/min. Along with the continuous isotope infusion the investigator will begin infusion of the Na-lactate at approximately 2.6mg/kg·min. Based upon readings from blood samples during the infusion, this rate will be adjusted as needed to maintain the target lactate concentration of approximately 4-5 mM. Blood samples will be drawn at 10, 20, 30, 45, 60, 75, 90 and 120 minutes, while breath samples will be collected at 60, 75, 90 and 120 minutes.
  Interventions: Other: Lactate infusion

INTERVENTIONS:
Other: Lactate infusion — The unlabeled lactate infusion cocktail (30% L(+)-lactic acid solution (Sigma) with 2N NaOH, pH4.8) and stable isotope infusions were made by a pharmacy and tested to be sterile and pyrogen free. Upon arriving to the KU Clinical and Translational Science Unit, a catheter will be placed in the subject's hand, which will be placed into a heated hand box for collection of arterialized blood. A second catheter will be placed in the opposing forearm vein for the infusion of lactate isotope solution and unlabeled lactate infusion cocktail. After insertion of the catheters, and prior to isotope infusion, a background blood and breath sample (ParvoMedics TrueOne 2400) will be obtained. We will then administer priming doses of 57.5 mg [13C3]lactate, 250 mg D2-glucose and 136 mg H13CO3- followed by continuous infusions of [13C3]lactate at 10 mg/min and D2-glucose at 2 mg/min [53]. Along with the continuous isotope infusion we will begin infusion of the Na-lact

SUMMARY:
Improved cardiorespiratory fitness following an aerobic exercise program elicits cognitive benefit in elderly subjects and memory improvement in Alzheimer's disease (AD). The physiological mechanism may be related to exercise-mediated change in circulating factors that permeate the brain. The response to each individual bout of exercise (i.e. the acute exercise response) may differ between subjects and be key to driving brain benefit. In young populations, the acute response to exercise can last hours and affect brain glucose metabolism. However, the field knows little about this acute exercise response in AD. Most exercise intervention trials designed to prevent and slow AD assess biomarkers at two fasting time points: pre- and post-intervention. The acute exercise response in the brain and periphery likely varies between subjects and diagnoses and provide key information regarding mechanisms of benefit. Our primary goals are to characterize the acute exercise response to exercise in the brain (glucose metabolism) and periphery (biomarker response) in aging and AD. We will identify relationships between exercise-related factors (i.e. heart rate, biomarkers) and change in brain metabolism and cognition. Understanding these mechanistic relationships will provide specific targets that can be used in future trials to develop individualized exercise prescriptions and maximize benefit.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common neurodegenerative disease, affecting over 5 million Americans, with this number expected to balloon to nearly 14 million by 2050. Annual health care costs associated with AD exceed 200 billion dollars which has led to the formation National Alzheimer's Project Act (NAPA). Goals of NAPA include the creation of a national plan to overcome AD, development of treatments to prevent, halt, or reverse AD, and improvements in early diagnosis and care of AD patients.

We have shown that an exercise program improves cognitive (primarily executive) function in cognitively healthy subjects in an exercise dose-dependent manner as well as a positive relationship between cardiorespiratory fitness change and memory change in individuals with AD who participate in 6 months of aerobic exercise. However, not all individuals benefit from exercise, and the precise mechanisms by which exercise elicits a beneficial effect are unclear. Most clinical trials, including our own, have been designed to assess metabolic outcomes at two fasting timepoints, before and after the intervention. However, the effects of each acute exercise bout on brain metabolism, and potential mechanisms by which cognition and memory may be affected, remain unclear. Longitudinal observational studies show a relationship between self-reported exercise and cognitive decline, and higher physical activity in midlife and late life is associated with a reduced risk of developing late-onset AD. Furthermore, intervention studies have shown cognitive improvement following exercise in ND and MCI subjects. Cardiorespiratory fitness decline tracks with brain atrophy and progression of dementia severity in AD and hippocampal volume has improved with a physical activity intervention in some studies of older adults. The fact that cardiorespiratory fitness change is important in achieving memory effects in AD is consistent with work that shows a positive relationship between exercise-related cardiorespiratory fitness change and markers of cortical thickness and brain volume in ND, MCI, and AD subjects. It is also consistent with work that shows physical activity and fitness levels are associated with larger brain volume. Cardiorespiratory fitness change is likely driven by the repeated, acute effects of each single, acute exercise bout that is additive over time. These acute effects include changes in peripheral biomarkers that readily cross the blood brain barrier but return to normal within a few hours. However, the effects of acute exercise on the brain are not well understood, especially in aged and AD populations, and at the intensities that are often used in exercise intervention programs. This presents a knowledge gap in the study of the beneficial effects of exercise in aging and dementia populations. One possible mediator of benefit with acute exercise is lactate. Production of lactate from pyruvate generates NAD+, a necessary intermediate for glycolysis. Peripheral lactate is transported to the liver for regeneration of pyruvate via the Cori cycle; however, lactate is transported throughout the entire body, and during physical exercise, lactate provides a key source of energy for muscle and brain. Lactate is used efficiently by the brain even at rest, the investigator hypothesize that lactate is a critical energy source for the brain, and that generation of lactate during acute exercise directly impacts glucose metabolism in the brain. This study will explore the effects of acute exercise on brain glucose metabolism as well as the dynamics of acute exercise biomarkers, including lactate and related substances that may affect brain metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older
* Stable medication doses (>1month)
* Post-menopausal
* Diagnosis of either Nondemented (CDR 0) or Probable AD (CDR 0.5 or 1 only)

Exclusion Criteria:

* Inability to provide consent
* Diagnosis of insulin-dependent (Type 1) Diabetes Mellitus
* Anti-platelet medication (Plavix), Warfarin, and other anticoagulants (Eliquis, Pradaxa, and Xarelto)
* Recent ischemic heart disease (<2 years)
* Diagnosis of a clinically significant chronic disease including CVD, other metabolic diseases (e.g., thyroid), cancer, HIV, or acquired immunodeficiency syndrome
* Any Neurological disorders that have the potential to impair cognition or brain metabolism (e.g., Parkinson's disease, stroke defined as a clinical episode with neuroimaging evidence in an appropriate area to explain the symptoms).
* Clinically significant depressive symptoms that may impair cognition, abnormalities in B12, RPR, or thyroid function that may impair cognition, use of psychoactive and investigational medications, and significant visual or auditory impairment

Ages: 60 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigator will leverage the KU ADC Outreach and Recruitment (OR) Core, which reaches more than 2000 individuals annually. The OR Core supports and maintains Eligibility Database, which contains demogrpahic and health information for all individuals who contact the ADC or are referred from clinic (n>7000, ~5000 without cognitive complaints). Recruitment will also leverage the ADC Clinical Cohort, which is comprised of 400 individuals who are characterized annually with clinical and cognitive testing.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Metabolic Clearance Rate (MCR) | 2 hours
  units of lactate cleared per minute (mg/kg×min)

SECONDARY OUTCOMES:
Cognitive Performace | 2 hours
  Calculate change in global cognition composite score between fasting and lactate-infused states

CONTACTS AND LOCATIONS:
Overall Officials: Jill Morris, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Univeristy of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kemna RE, Kueck PJ, Blankenship AE, John CS, Johnson CN, Green ZD, Chamberlain T, Thyfault JP, Mahnken JD, Miller BF, Morris JK. Methods to characterize lactate turnover in aging and Alzheimer's disease; The LEAN study. Contemp Clin Trials. 2024 Nov;146:107682. doi: 10.1016/j.cct.2024.107682. Epub 2024 Sep 3. PMID 39236780